CLINICAL TRIAL: NCT01918527
Title: Neoadjuvant Chemotherapy Versus Standard Treatment in Patients With Locally Advanced Colon Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoCol
Record Dates: First submitted 2013-08-06; First posted 2013-08-07 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Colon Cancer
Keywords: Locally advanced colon cancer; Neoadjuvant chemotherapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A, Conventional treatment (Other): Operation + 4 or 8 cycles of adjuvant chemotherapy, if indicated.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin
- B, Neoadjuvant chemotherapy (Other): 3 cycles of neoadjuvant chemotherapy + operation. Adjuvant chemotherapy only if indicated.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine — Orally on days 1-14: 2000 mg/m2/day q3w
Drug: Oxaliplatin — Intravenously on day 1: 130 mg/m2 q3w

SUMMARY:
The purpose of this study is to compare 3 cycles of neoadjuvant (preoperative) chemotherapy + operation with the standard treatment of locally advanced colon cancer, which is operation + 8 cycles of (adjuvant) chemotherapy.

Patients receiving neoadjuvant chemotherapy may not need adjuvant chemotherapy after the operation and, if this is the case, they will be spared of 5 cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified locally advanced T3 (ETI > 5 mm) or T4 colon cancer assessed by CT scan.
* Age ≥ 18 years
* PS 0-2.
* Hematology ANC ≥1.5x10^9/l. Thrombocytes ≥ 100x10^9/l.
* Biochemistry Bilirubinemia ≤ 3 x upper normal level. ALAT ≤ 5 x upper normal value
* Consent to translational research
* Fertile women must present a negative pregnancy test and use secure contraceptives during and 3 months after treatment.
* Written and orally informed consent.

Exclusion Criteria:

* Patients with distant metastases.
* Acute operation
* Clinically significant cardiovascular disease (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before inclusion.
* Active, serious infection or other serious disease.
* Peripheral neuropathy NCI grade > 1
* Other malignant disease within 5 years prior to study enrollment, except basocellular or squamous skin cancer and carcinoma in situ cervicis uteri.
* Other investigational treatment within 30 days prior to treatment start.
* Hypersensitivity to one or more of the active or auxiliary substances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Two-year disease free survival | 2 years after completed study treatment

SECONDARY OUTCOMES:
Rate of patients fulfilling the criteria for adjuvant chemotherapy | 6, 12, 18, and 24 months after completed study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jakobsen, DMSc, Study Chair — Vejle Hospital, Vejle, Denmark; Henrik Jensen, MD, PhD, Principal Investigator — Vejle Hospital, Vejle, Denmark; Olav Dahl, MD, Principal Investigator — Haukeland University Hospital, Bergen, Norway; Göran Carlsson, MD, Principal Investigator — Sahlgrenska University Hospital
Locations (9):
- Denmark (7):
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Hilleroed Hospital, Hillerød
  - Roskilde Hospital, Roskilde
  - Sygehus Sønderjylland, Sønderborg
  - Vejle Hospital, Vejle
- Haukeland University Hospital, Bergen, Norway
- Sahlgrenska University Hospital, Gothenburg, Sweden